CLINICAL TRIAL: NCT05983263
Title: Neuropathic Determining Factors and Analgesic Efficacy of Capsaicin 8% (QUTENZA®) Patches in Refractory Coccygodygnia
Brief Title: Analgesic Efficacy of Capsaicin 8% Patch (QUTENZA®) in Coccygodygnia
Acronym: CAPSACOXp
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CAPSACOXp_AL_06032023
Record Dates: First submitted 2023-03-06; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Coccyx Disorder
Keywords: Chronic Coccygodynia; Neuropathic pain; Capsaicine 8%
MeSH Terms: conditions — Neuralgia | interventions — Capsaicin; Transdermal Patch

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Capsaicin — Capsaicin 8% patch (QUTENZA) apposed in coccygeal area
  Other Names: Capsaicin 8% patch

SUMMARY:
A retrospective study over a period of 6 years to explore analgesic efficacy of 8% Capsaicin patch (QUTENZA®) in coccygodynic patients, as well as neuropathic predictive factors of therapeutic response.

DETAILED DESCRIPTION:
Coccygodynia corresponds to a localized pain in the coccyx region, aggravated or triggered by sitting and/or by getting up from a seat. Even if there is no epidemiology of this pain in France, coccygodynia represents a frequent recourse to specialized consultations (Rheumatology or Algology). Currently in France, there is no recommendation on the management of chronic disabling coccygodynia. Treatments are proposed in accordance with known/presumed underlying pathophysiology. Anti-inflammatory drugs and manual therapy (pressure relief cushions) are thus always offered as first-line treatments. But despite their common use/prescription, their efficacy is variable, with low level of evidence. More over, upstream of invasive coccygectomy, therapeutic arsenal is largely deficient, inviting to explore new approaches. Considering frequent neuropathic expression in coccygodynic pain pattern (tingling, itching, pain cold sensation…), capsaïcine 8% patch (QUTENZA®) are often performed. And in the same way, no/few researches tried to measure real-life analgesic pain efficacy of QUTENZA® strategy. Observational retrospective study (non-interventional anonymized data) CAPSACOXp aims to assess analgesic efficacy of Capsaicin 8% patch (QUTENZA®) and explore possible neuropathic determinants of therapeutic response in coccygodynia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received topical Capsaicin 8% patch therapy for the treatment of their coccygodygnia between August 2016 and August 2022

Exclusion Criteria:

* Patients who have already received 8% Capsaicin patch topical treatment in coccyx area.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical files of 106 patients hospitalized between 2016 and 2022 for persisting coccygodynia (>3months) and at least one neuropathic symptom in pain expression, and who received capsaicin 8% patch (QUTENZA®) topical treatment.
Sampling Method: Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2023-12-17 (Estimated); Study Completion 2023-12-21 (Estimated)

PRIMARY OUTCOMES:
Responder rate | 3 months after the inclusion visit.
  Success defined by PGIC ≤ 2.

SECONDARY OUTCOMES:
Therapeutic response neuropathic predictive factors | 3 months after the inclusion visit
  Identification of baseline neuropathic predictive factors (extracted from DN4 criteria) of Capsaïcine 8% efficacy at 3months (ie. PGIC ≤ 2)

IPD SHARING:
Plan to Share IPD: No
Anonymized dataset. No sharing.